CLINICAL TRIAL: NCT06747182
Title: Mobile Phone-based Smoking Cessation Program for Individuals With Cardiovascular Risk or Disease in China
Brief Title: Mobile Phone-based Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0716
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2023-04

CONDITIONS: Substance Use Disorder (SUD)
Keywords: smoke cessation; cardiovascular diseases
MeSH Terms: conditions — Substance-Related Disorders; Smoking Cessation; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the wait-list control group (No Intervention): the wait-list control group
- mobile phone-based intervention group (Experimental): Participants will receive a 12-week intervention with follow-up at week 26.
  Interventions: Other: mobile phone-based intervention

INTERVENTIONS:
Other: mobile phone-based intervention — Participants in intervention group will receive a 12-week mobile phone-based intervention with follow-up at week 26.
  Arms: mobile phone-based intervention group

SUMMARY:
In this online, randomized controlled trial (RCT), the participants will be randomized and allocated in 1:1 ratio to mobile phone-based intervention group or to the wait-list control group. Participants will receive a 12-week intervention with follow-up at week 26. The primary outcome includes biologically verified continuous smoking abstinence at week 26 after the quit date. The main secondary outcomes include seven-day point prevalence smoking abstinence at weeks 1, 2, 3, 4, 8, 12, 16, 20 and 26, self-reported continuous smoking abstinence at weeks 4, 8, 12, 16, 20 and 26 after the quit date. About 2000 smokers with willingness to make a quit attempt within a month from October 2022 to April 2023 or until the recruitment process is complete will be recruited. The final 26-week follow-up will be completed in November 2023. The trial results will be available by the end of 2023 .

ELIGIBILITY:
Inclusion Criteria:

* In this RCT, approximately 2,000 smokers (a smoker is defined as an individual who smoked 100 cigarettes in their lifetime, and currently smoke ≥ 5 cigarettes per day) who are willing to make a quit attempt within one month with CVDs diagnosis or risk.

Exclusion Criteria:

* patients unwilling to quit smoking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Continuous smoking abstinence | at week 26 after the quit date
  biologically verified continuous smoking abstinence at week 26 after the quit date

SECONDARY OUTCOMES:
7-day point prevalence smoking abstinence | week 1, 2, 3, 4, 8, 12, 16, 20 and 26
  seven-day point prevalence smoking abstinence at weeks 1, 2, 3, 4, 8, 12, 16, 20 and 26
self-reported continuous smoking abstinence | week 4, 8, 12, 16, 20 and 26 after the quit date
  self-reported continuous smoking abstinence at weeks 4, 8, 12, 16, 20 and 26 after the quit date

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, China., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No